CLINICAL TRIAL: NCT00136929
Title: A Prospective Randomized Trial of Primary Angioplasty Versus Thrombolytic Therapy for Acute Myocardial Infarction in the Elderly "Senior PAMI"
Brief Title: Senior PAMI: Primary Angioplasty Versus Thrombolytic Therapy for Acute Myocardial Infarction in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PAMI Coordinating Center (Other)
Collaborators: Eli Lilly and Company (Industry); Guidant Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC 1999-225
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2005-08

CONDITIONS: Myocardial Infarction
Keywords: AMI; MI; Acute myocardial infarction (AMI), (MI)
MeSH Terms: conditions — Myocardial Infarction | interventions — Thrombolytic Therapy; Percutaneous Coronary Intervention

INTERVENTIONS:
Drug: Thrombolytic therapy
Procedure: Percutaneous coronary intervention (PCI)

SUMMARY:
This is a prospective, randomized, multi-center, international trial comparing two reperfusion strategies in elderly (age >= 70 years) patients with acute myocardial infarction: primary percutaneous coronary intervention (PCI) versus intravenous thrombolytic therapy. Clinical endpoints will be collected in the hospital, at 1 month, 6 months, and 1 year post-randomization. The primary endpoint is 30 day death or disabling stroke. The study null hypothesis is that there will be no significant difference in death or disabling stroke at 30 days post-randomization between patients treated with PCI versus thrombolytics.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 70
* Clinical symptoms > 30 minutes
* Symptom onset <= 12 hours
* ST segment elevation >= 1 mm in 2 or more leads

Exclusion Criteria:

* Prior thrombolytics
* Cardiogenic shock
* Cerebrovascular accident (CVA)
* Prolonged cardiopulmonary resuscitation (CPR)
* Blood pressure (BP) > 180/100 mm Hg
* Active bleeding
* International Normalized Ratio (INR) > 1.4
* Acetylsalicylic acid [aspirin] (ASA) or heparin allergy
* History of neutropenia, thrombocytopenia, hepatic dysfunction, or renal insufficiency
* Peripheral vascular disease (PVD)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 530

CONTACTS AND LOCATIONS:
Overall Officials: Felix Zijlstra, M.D., Principal Investigator — Ziekenhuis de Weezenlanden